CLINICAL TRIAL: NCT01668173
Title: A Phase II Study of the HSP90 Inhibitor, AUY922, in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF), and Refractory PV/ET
Brief Title: HSP90 Inhibitor, AUY922, in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF), and Refractory PV/ET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: patient safety
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-076
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Myeloproliferative Neoplasms
Keywords: HSP90 Inhibitor; AUY922; 12-076
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

ARMS (1):
- AUY922 (Experimental): This is an open-label phase II trial to assess the efficacy of the HSP90 inhibitor, AUY922, in patients with PMF, post-PV MF, post-ET MF, and with PV/ET who are refractory to hydroxyurea, phlebotomy or anagrelide.
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY922 will be administered as an intravenous infusion over 60 minutes, on a once weekly schedule. A cycle on study will be defined as 28 days. The dose to be studied are 70 mg/m2 and 55 mg/m2 if DLTs are identified in the first 3-6 patients. The same schedule of administration will be used for all patients in this trial.

SUMMARY:
The purpose of this study is to test a new drug called AUY922. AUY922 is not FDA-approved. AUY922 is a new kind of drug that attacks a protein called HSP90. HSP90 is found in both normal and cancer cells, but the investigators think it is more important in cancer cells.

This study will see if AUY922 helps people with myelofibrosis, essential thrombocythemia and polycythemia vera. This study will also see if AUY922 is safe in people with myelofibrosis, essential thrombocythemia and polycythemia vera. It will find out what effects, good and/or bad, AUY922 has on the patient and the disease. The researchers hope that this study will help them to find better treatments for primary myelofibrosis, essential thrombocythemia and polycythemia vera.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have myeloproliferative neoplasms, specifically, primary myelofibrosis (PMF), post polycythemia vera myelofibrosis (post-PV MF), post essential thrombocythemia myelofibrosis (post-ET MF), and PV/ET that are refractory to hydroxyurea, phlebotomy and anagrelide or not a candidate for standard therapies.
* ≥ 18 years of age
* ECOG performance status of 0-2
* Acceptable pre-study organ function during screening as defined as:

Hematologic:

* Absolute Neutrophil Count (ANC) ≥1.5x109/L
* Hemoglobin (Hgb) ≥ 8 g/dl (may be supported with transfusion)
* Platelets (plt) ≥50x10^9/L

Biochemistry:

* Potassium within normal limits
* Total calcium (corrected for serum albumin) and phosphorus within normal limits
* Magnesium above LLN or correctable with supplements Liver and Kidney Functions
* AST/SGOT and ALT/SGPT ≤ 1.5 x Upper Limit of Normal (ULN) if AP > 2.5 X ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5
* Serum bilirubin ≤ 1.5 x ULN (Unless attributable to Gilbert's disease)
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 ml/min
* Negative serum pregnancy test. The serum pregnancy test must be obtained prior to the first administration of AUY922 (≤ 72 hours prior to dosing) in all pre-menopausal women and women <2 years after the onset of menopause
* Patients who previously received JAK2 inhibitors will be eligible as long as they have been off the drug for more than 4 weeks.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Requiring ongoing therapy with either G- or GM-CSF, or long-acting versions of these molecules
* Active medical condition such as infection or cancer that is actively requiring treatment.
* Unresolved diarrhea ≥ CTCAE (v4.02) grade 1
* Prior anti-neoplastic treatment with any HSP90 or HDAC inhibitor compound
* Patients who have undergone any major surgery ≤ 2 weeks prior to starting study drug or have not recovered from the side effects of such therapy.
* Patient must be ≥ 4 weeks since last chemotherapy or treatment with another systemic anticancer agent with the exception of hydroxyurea. Hydroxyurea must be discontinued at least 48 hours prior to the initiation of AUY922. Patients must have recovered (CTC ≤ 1) from acute toxicities of any previous therapy (with the exception of alopecia).
* Active anticoagulation with warfarin.
* Pregnant or lactating women
* Fertile women of childbearing potential (WCBP) not using double-barrier methods of contraception (abstinence, oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly, or surgically sterile). Male patients whose partners are WCBP not using double-barrier methods of contraception.

Impaired cardiac function, including any one of the following:

* History (or family history) of long QT syndrome
* Mean QTc ≥ 450 msec on baseline ECG
* History of clinically manifested ischemic heart disease (including myocardial infarction, stable or unstable angina pectoris, coronary arteriography or cardiac stress testing/imaging with findings consistent with infarction or clinically significant coronary occlusion) ≤ 6 months prior to study start
* History of heart failure or left ventricular (LV) dysfunction (LVEF ≤ 45%) by MUGA or ECHO
* Clinically significant ECG abnormalities including 1 or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB). ST segment elevation or depression > 1mm, or 2nd (Mobitz II), or 3rd degree AV block.

History or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes

* Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Clinically significant resting bradycardia (< 50 beats per minute)
* Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the QTcF interval or inducing Torsades de Pointes and cannot be switched or discontinued to an alternative drug prior to commencing AUY922.
* Obligate use of a cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raajit Rampal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: HSP90 Inhibitor, AUY922, in Patients with Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), Post-Essential Thrombocythemia Myelofibrosis (Post-ET MF), and Refractory PV/ET
Period: Overall Study
Arm/Group | All Patients
Started | 7
Completed | 0
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Trial suspension | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Number; unit: participant with Stable Disease
Arm/Group | All Patients
Number analyzed (Participants) | 1
participant with Stable Disease | 1

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=7)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ileal ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=7)
Pain (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Anorexia (General disorders) | 1
Bloating (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Insomnia (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Back pain (General disorders) | 1
Bone pain (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5
CPK increased (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Rash pustular (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (General disorders) | 2
Blurred vision (General disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Night blindness (General disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Lipase increased (Metabolism and nutrition disorders) | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Creatinine increased (Metabolism and nutrition disorders) | 2
Serum amylase increased (Metabolism and nutrition disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 2
Blood bilirubin increased (Metabolism and nutrition disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Psychiatric disorders - Other (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes